CLINICAL TRIAL: NCT07160257
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Maridebart Cafraglutide on Insulin Sensitivity and β-cell Function in Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of Maridebart Cafraglutide on Insulin Sensitivity and β-cell Function in Participants With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20250061
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; T2DM; Maridebart Cafraglutide; AMG 133; Insulin sensitivity; β-cell Function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maridebart cafraglutide (Experimental): Participants will receive maridebart cafraglutide subcutaneously (SC).
  Interventions: Drug: Maridebart cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart cafraglutide — Maridebart cafraglutide will be administered SC.
  Other Names: AMG 133
  Arms: Maridebart cafraglutide
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effect of maridebart cafraglutide relative to placebo on insulin sensitivity in participants with Type 2 Diabetes Mellitus (T2DM) treated with stable dose of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent before initiation of any study-specific activities/procedures.
* Male or female participants aged ≥ 18 and ≤ 70 years at the time of signing informed consent.
* Body mass index 27 ≥ and ≤ 45 kg/m^2 at screening.
* Diagnosis of T2DM at least 6 months before screening based on the WHO classification.
* Treatment of T2DM for at least 3 months prior to screening with diet and exercise and a stable dose of metformin (either immediate release or extended release), with or without a stable dose of 1 additional OAM other than metformin.

Exclusion Criteria:

* Type 1 diabetes mellitus, history of ketoacidosis or hyperosmolar state/coma, or any other type of diabetes mellitus (except T2DM or history of gestational diabetes).
* History of proliferative diabetic retinopathy or diabetic macular edema or nonproliferative diabetic retinopathy that requires acute treatment.
* One or more episodes of severe hypoglycemia (Level 3 hypoglycemia as defined by the American Diabetes Association classification criteria) within 6 months before screening, as defined by the occurrence of neuroglycopenic symptoms requiring the assistance of another person for recovery.
* Has modified diet or adopted any nutritional lifestyle modifications within 3 months prior to screening, as assessed by the investigator (or designee) based on participant self-report.
* History of malignancy within the last 5 years before screening (except nonmelanoma skin cancers, cervical carcinoma in situ, or breast ductal carcinoma in situ).
* Family (first-degree relative[s]) or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN-2).
* History or evidence of endocrine disorder (such as Cushing's syndrome) that can cause obesity.
* History or evidence of autoimmune disease that can directly or indirectly affect insulin production, insulin action, or glucose metabolism.
* History of any of the following within 90 days before screening: myocardial infarction, unstable angina, coronary artery bypass graft surgery or other major cardiovascular surgery, percutaneous coronary intervention (diagnostic angiograms are permitted), transient ischemic attack, cerebrovascular accident, or decompensated congestive heart failure, or currently have New York Heart Association Class III or IV heart failure.
* History of chronic pancreatitis.
* History of acute pancreatitis within 6 months before screening.
* Positive human immunodeficiency virus test at screening.
* Evidence of hepatitis B or C infection.
* Estimated glomerular filtration rate < 60 mL/min/1.73 m^2 calculated by the 2021 Chronic Kidney Disease Epidemiology Collaboration creatinine-cystatin C equation at screening.
* Hemoglobin value < 12 g/dL (males) or < 10 g/dL (females) at screening or check-in (Day -4).
* Use within 90 days before randomization of medications, supplements, or alternative remedies for weight loss (eg, GLP-1RA, GIP agonists, phentermine/topiramate, naltrexone/bupropion, orlistat, and sympathomimetic drugs).
* Use within 90 days before randomization of chronic (> 14 days) systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, intraarticular, or inhaled preparations).
* Use within 90 days before randomization of medications that may cause significant weight gain including, but not limited to, atypical antipsychotic and mood stabilizers.
* Current or prior use of herbal supplements that affect insulin or glucose within 30 days before randomization.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days (or 5 half-lives, whichever is longer) since ending treatment on another investigational device or drug study(ies).
* Participants of childbearing potential unwilling to adhere to contraception requirements during treatment and for an additional 16 weeks after the last dose of IMP.
* Participants who are breastfeeding or who plan to breastfeed while on study through 16 weeks after the last dose of IMP.
* Participants planning to become pregnant while on study through 16 weeks after the last dose of IMP.
* Major surgical procedure planned during the study.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease (except for those outlined above) that, in the opinion of the investigator or medical monitor, if consulted as necessary, would pose a risk to participant's safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in M-value from Hyperinsulinemic-euglycemic Clamp at Week 25 | Baseline and Week 25

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events and Serious Adverse Events | Up to Week 41
Plasma Concentration of Maridebart Cafraglutide at Week 25 | Week 25
Number of Participants with Anti-maridebart Cafraglutide Antibody Formation | Up to Week 41
Change from Baseline in Total Insulin Secretion at Week 25 | Baseline and Week 25
  Measured as area under the curve (AUC) of insulin secretion rate (ISR) from hyperglycemic clamp (ISR0-120min).
Change from Baseline in First Phase Incremental ISR from Hyperglycemic Clamp (ISR0-8min) at Week 25 | Baseline and Week 25
Change from Baseline in Second Phase Insulin Secretion at Week 25 | Baseline and Week 25
  Measured as AUC of ISR from hyperglycemic clamp (ISR20-120min).
Change from Baseline in Maximum Insulin Secretion at 8 Minutes at Week 25 | Baseline and Week 25
  Measured as incremental ISR responses to arginine from hyperglycemic clamp at 8 minutes (ISRarg0-8min).
Change from Baseline in Maximum Insulin Secretion at 30 Minutes at Week 25 | Baseline and Week 25
  Measured as incremental ISR responses to arginine from hyperglycemic clamp at 30 minutes (ISRarg0-30min).
Change from Baseline in ISR at Week 25 | Baseline and Week 25
  Measured as total AUC (ISR0-240min) from standardized mixed meal tolerance test (sMMTT).
Change from Baseline in Clamp Disposition Index (cDI) at Week 25 | Baseline and Week 25
  Calculated as product of M-value and ISR0-120min from the hyperglycemic clamp.
Change from Baseline in Post-meal Glucose Concentrations During sMMTT (Total and Incremental AUC0-240min) at Week 25 | Baseline and Week 25
Change from Baseline in Hemoglobin A1c (HbA1c) at Week 25 | Baseline and Week 25
Change from Baseline in Fasting Glucose Concentration at Week 25 | Baseline and Week 25
Change from Baseline in Fasting Glucagon Concentration at Week 25 | Baseline and Week 25
Change from Baseline in Glucagon Concentration During sMMTT (Total and Incremental AUC0-240min) at Week 25 | Baseline and Week 25
Change from Baseline in Fasting Triglycerides at Week 25 | Baseline and Week 25
Change from Baseline in Fasting High-density Lipoprotein-cholesterol (HDL-C) at Week 25 | Baseline and Week 25
Change from Baseline in Fasting Non-HDL-C at Week 25 | Baseline and Week 25
Change from Baseline in Triglyceride Concentration During sMMTT (Total and Incremental AUC0-240min) at Week 25 | Baseline and Week 25
Change from Baseline in Fasting Free Fatty Acids (FFA) Concentration (During Hyperinsulinemic-euglycemic Clamp and sMMTT) at Week 25 | Baseline and Week 25
Change from Baseline in FFA Concentrations During sMMTT (Total AUC0-240min) at Week 25 | Baseline and Week 25
Change from Baseline in Percentage Body Fat at Week 25 | Baseline and Week 25
Change from Baseline in Body Fat Mass at Week 25 | Baseline and Week 25
Change from Baseline in Lean Body Mass at Week 25 | Baseline and Week 25
Change from Baseline in Body Weight at Week 25 | Baseline and Week 25
Change from Baseline in Waist Circumference at Week 25 | Baseline and Week 25
Change from Baseline in Hunger Fasting Appetite Visual Analog Scale (VAS) Score at Week 25 | Baseline and Week 25
Change from Baseline in Satiety Fasting Appetite VAS Score at Week 25 | Baseline and Week 25
Change from Baseline in Fullness Fasting Appetite VAS Score at Week 25 | Baseline and Week 25
Change from Baseline in Prospective Food Consumption Fasting Appetite VAS Score at Week 25 | Baseline and Week 25
Change from Baseline in Overall Fasting Appetite VAS Score at Week 25 | Baseline and Week 25
Change from Baseline in Hunger Appetite VAS Score During sMMTT at Week 25 | Baseline and Week 25
Change from Baseline in Satiety Appetite VAS Score During sMMTT at Week 25 | Baseline and Week 25
Change from Baseline in Fullness Appetite VAS Score During sMMTT at Week 25 | Baseline and Week 25
Change from Baseline in Prospective Food Consumption Appetite VAS Score During sMMTT at Week 25 | Baseline and Week 25
Change from Baseline in Overall Appetite VAS Score During sMMTT at Week 25 | Baseline and Week 25
Change from Baseline in Food Craving Inventory (FCI) Score at Week 25 | Baseline and Week 25
Change from Baseline in Caloric Intake During Ad Libitum Meal at Week 25 | Baseline and Week 25

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- ProSciento, Inc. - Main Clinic, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com